CLINICAL TRIAL: NCT05507411
Title: Watch and Wait for NeoAdjuvant Concurrent Radiochemotherapy Combined With Camrelizumab in Patients With Resectable Esophageal Squamous Cell Carcinoma，A Prospective, Single-Center, Open Label，Phase II Cohort Study （WATCHER）
Brief Title: Watch and Wait for NeoAdjuvant Concurrent Radiochemotherapy Combined With Camrelizumab in Patients With Resectable ESCC
Acronym: WATCHER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Qixun Chen, Director, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WATCHER
Record Dates: First submitted 2022-08-12; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; NeoAdjuvant therapy; immunotherapy; Concurrent Radiochemotherapy; organ preservation
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CCR-Watch and Wait (Other)
  Interventions: Radiation: Neoadjuvant Radiotherapy; Drug: Neoadjuvant Chemotherapy; Drug: Immunotherapy
- CCR-Surgery (Other)
  Interventions: Radiation: Neoadjuvant Radiotherapy; Drug: Neoadjuvant Chemotherapy; Drug: Immunotherapy
- Non-CCR (Other)
  Interventions: Radiation: Neoadjuvant Radiotherapy; Drug: Neoadjuvant Chemotherapy; Drug: Immunotherapy

INTERVENTIONS:
Radiation: Neoadjuvant Radiotherapy — 41.4Gy/23F
Drug: Neoadjuvant Chemotherapy — Paclitaxel for Injection （Albumin Bound): 50mg/m^2 QW Carboplatin: AUC=2 QW
Drug: Immunotherapy — Camrelizumab 200mg Q3W

SUMMARY:
To observe the 1-year disease-free survival rate （1-year PFS） of patients with resectable esophageal squamous cell carcinoma who received neoadjuvant chemoradiotherapy combined with camrelizumab and achieved clinical complete remission with watchful waiting strategy.

DETAILED DESCRIPTION:
This trial is a prospective, multicenter, randomized controlled phase II clinical study.

Eligible patients with thoracic esophageal squamous cell carcinoma in clinical stage cT2-4aNanyM0, or cT1-3N+M0. The patient received radiotherapy (41.4Gy/23F), chemotherapy (nab-paclitaxel combined with carboplatin), immunotherapy (Camrelizumab), and a combination of imaging, endoscopy and biopsy pathology was performed 4-6 weeks after the end of neoadjuvant therapy.

Evaluate (CRE1) to determine whether clinical complete resection (cCR) has been achieved. If clinical complete resection is not reached, patients will receive radical surgery; For subjects who have achieved clinical complete resection（cCR）, they will be randomly divided into an operation group and an observational waiting group. After 14 weeks, the combined imaging, endoscopy and biopsy pathological evaluation (CRE2) was performed again to determine whether the clinical complete resection (CCR2) was reached. If the patient has local progression and can be resected, radical surgery will be performed; if there is distant progression, medical oncology treatment or supportive treatment will be performed; if clinical complete resection remains, continuous and close imaging, endoscopic and Biopsy pathology combined evaluation (CRE3-14). After achieving clinical complete resection, patients who continue to be followed up for observation or undergo radical surgery, if there is no contraindication to treatment, receive 14 cycles of Camrelizumab maintenance therapy. During follow-up stage, if the patient develops local progression and can be resected, radical surgery is performed; if distant progression occurs, medical oncology treatment or supportive treatment is performed; if clinical complete remission is still achieved, follow-up evaluation can be continued. Among them, the 1-year disease-free survival rate under the esophagus-sparing treatment strategy after achieving clinical complete remission was the main endpoint of the study.

To observe the disease-free survival（DFS）, overall survival（OS）, event-free survival（EFS）, quality of life（QoL）, failure mode and choice of post-failure treatment mode after neoadjuvant chemoradiotherapy combined with Camrelizumab therapy or after surgical resection. And, the pathological complete remission rate and the main pathological resection rate of the patients who underwent surgery.

The blood, stool and tissue samples of patients participating in the trial will be retained for future detection of relevant markers and related laboratory research.

Treatment safety and toxicity, including acute and chronic toxicity, will be evaluated on an ongoing basis during treatment and follow-up.

Any serious adverse drug reactions will be promptly reported to the hospital ethics committee.

The relationship between relevant markers and clinical outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent. Participants signed and dated written informed consent. Informed consent must be signed prior to any protocol-related procedures that are not part of the participant's routine medical care； Participants must be willing and able to comply with scheduled visits, treatment regimens, and laboratory tests；
2. Participant type and target disease characteristics Eastern Collaboration Group (ECOG) physical status score 0-1； Histologically confirmed esophageal cancer with lesions located in the thoracic esophagus, AJCC/UICC esophageal cancer staging (eighth edition) clinical stage cT2-4aNanyM0, or cT1-3N+M0； Presence of measurable lesions according to RECIST criteria； Participants must have tumor tissue samples available for PD-L1 IHC testing； No major associated pathological conditions that increase the risk of surgery to unacceptable levels. Such as: esophageal perforation and active esophageal bleeding, obvious trachea, thoracic large blood vessel invasion； According to the surgeon's assessment, the total lung function can withstand the proposed esophageal cancer resection；
3. Age and reproductive status Age ≥18 years old and ≤75 years old； Females of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity of 25 IU/L or equivalent for HCG) within 24 hours prior to initiation of study treatment； Women must be non-nursing；

Exclusion Criteria:

1) Medical condition There is locally advanced unresectable (regardless of stage) or metastatic disease.

Participants with Grade ≥2 Peripheral Neuropathy； Participants with active, known or suspected autoimmune disease. Participants with type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, skin disorders that do not require systemic treatment (eg, vitiligo, psoriasis, or alopecia), or disorders that are not expected to recur in the absence of external stimuli are eligible to be enrolled； Participants requiring systemic therapy with glucocorticoids (>10 mg prednisone equivalent daily) or other immuno suppressive drugs within 14 days prior to treatment. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal hormone replacement therapy at >10 mg prednisone-equivalent daily are permitted； Known history of positive human immuno deficiency virus (HIV) test or known acquired immuno deficiency syndrome (AIDS)； Participants with serious or uncontrolled medical illness； previous/concomitant therapy； Received chest radiotherapy, chemotherapy, immunotherapy, or surgery of the esophagus, esophagus and gastric junction, or stomach prior to the start of the trial.

Patients with severe cardiovascular or pulmonary disease, interstitial pneumonia, or previous history of interstitial pneumonia； Patients with obvious esophageal ulcers, moderate pain in the chest and back, and esophageal perforation symptoms； Physical examination and laboratory test results

Laboratory screening values must meet the following criteria (using CTCAE 4th edition):

i) WBC < 2000/μL； ii) Neutrophils < 1500/μL； iii) Platelets < 100x103/μL； iv) Hemoglobin < 9.0 g/dL； v) Serum creatinine <1.5 x ULN or calculated creatinine clearance (CrCl) < 50 mL/min (using Cockcroft-Gault formula)； vi) AST >3.0 x ULN； vii) ALT > 3.0 x ULN； viii) Total bilirubin >1.5 x ULN (except for Gilbert syndrome participants, who had total bilirubin < 3.0 x ULN)； Participants had active hepatitis B (positive for hepatitis B surface antigen [HBsAg] or positive for hepatitis C virus (HCV) (positive for HCV RNA)； i) Participants with previous or recovered HBV infection (defined as having hepatitis B core antibody [HBcAb] and no HBsAg) are eligible. HBV DNA from these patients must be obtained prior to treatment. Participants who are HBV carriers or require antiviral therapy are not eligible； ii) Participants positive for HCV antibodies are eligible only if PCR for HCV RNA is negative.； Active malignancy within the past 3 years, except for locally curable cancers that have been significantly cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast； Participants with serious or uncontrolled medical conditions； Allergic Reactions and Adverse Drug Reactions； History of allergic reactions or hypersensitivity reactions to study drug components Other exclusion criteria； Patients who do not understand trial requirements, or who may not comply with trial requirements； Active infection requiring systemic therapy 14 days prior to first dose Some obvious diseases that the researchers believe should be excluded from this study；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
1-year DFS of CCR-Watch and Wait group | 1 year

SECONDARY OUTCOMES:
Overall Survival | 5 years
EFS | 5 years
cCR rate | 1 year
pCR rate | 1 year
MPR rate | 1 year
FACT-E | 5 years
  Quality of life
EORTC QLQ-30 | 5 years
  Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Qixun Chen, Principal Investigator — Zhejiang Cancer Hospital; Yongling Ji, Principal Investigator — Zhejiang Cancer Hospital
Locations (3):
- China (3):
  - The First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hanzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hanzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Batran SE, Koch C. Neoadjuvant therapy for oesophageal cancer: refining the armamentarium. Lancet. 2024 Jul 6;404(10447):5-7. doi: 10.1016/S0140-6736(24)01084-5. Epub 2024 Jun 11. No abstract available. PMID 38876135